CLINICAL TRIAL: NCT02440737
Title: Navigated Early Survivorship Transition in Improving Survivorship Care Planning in Patients With Newly Diagnosed Cancer and Their Caregivers (NEST)
Brief Title: Navigated Early Survivorship Transition in Patients With Newly Diagnosed Cancer and Their Caregivers
Acronym: NEST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Debra Friedman, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VICC REACH 1525; NCI-2015-00470 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); VICC REACH 1525 (Other: VICC (Vanderbilt Ingram Cancer Center)); P30CA068485 (NIH)
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Cancer
Keywords: Newly diagnosed; Cancer patient; Caregiver; Support person
MeSH Terms: conditions — Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods; Aftercare; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NEST Intervention (Experimental): Patients (PTs) and their caregivers (CGs) receive educational intervention, follow-up care, psychosocial assessment and care, and questionnaire administration interventions by completing psychosocial questionnaires and meeting with a nurse practitioner (NP) or nurse navigator (NN) for an initial survivorship care planning session to review the expected course of therapy and recovery, identify resources that may be needed and provide recommendations for follow-up. At the end of their treatment EOT), PTs and their CGs complete a 2nd set of questionnaires and meet with the NP/NN for a booster survivorship care planning session. They will receive an individualized final survivorship care plan and related materials. 2 months after EOT, PTs and their CGs complete a final set of questionnaires.
  Interventions: Other: Educational Intervention; Other: Follow-Up Care; Procedure: Psychosocial Assessment and Care; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Receive publication, "When Someone You Love is Being Treated for Cancer", a preliminary individualized Survivorship Care Plan (SCP), a final individualized SCP, and the "REACH for Survivorship" handbook.
  Other Names: Education for Intervention; Intervention, Educational
Other: Follow-Up Care — Complete Survivorship Care Planning session at end of treatment
Procedure: Psychosocial Assessment and Care — Undergo the NEST intervention
  Other Names: Psychosocial Assessment; Psychosocial Care; Psychosocial Care/Assessment; Psychosocial Studies; Psychosocial Support
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies the Navigated Early Survivorship Transition (NEST) intervention in improving survivorship care planning in patients with newly diagnosed cancer and their caregivers. A survivorship care planning session (SCPS) delivered to survivors and their primary caregivers may improve psychosocial well-being, patient and caregiver engagement, and adherence to treatment and follow-up recommendations. It is not yet known whether a NEST intervention or usual care is better in improving survivorship care planning in patients with newly diagnosed cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. In a new model of survivorship care planning, planning started within the first two months of therapy, followed by additional survivorship care planning at the end of therapy or 6 months post diagnosis, evaluate the proportion of eligible survivors and participating caregivers who complete the survivorship care planning.

II. In a feasibility study of survivors and their identified support caregivers (70 survivors with or with a participating caregiver at VICC and 70 survivors with or without a participating caregiver at MMC), evaluate psychosocial well-being, engagement, resource utilization and adherence to recommended treatment and follow-up guidelines.

III. Assess the outcomes of survivors and participating caregivers treated at VICC and MMC to further individualize survivorship planning that will incorporate the optimal timing and content together with socioeconomic and cultural considerations. The pillars of this novel intervention (i.e., survivorship care planning, psychosocial assessment and patient engagement) are responsive to the recommendations of the IOM. The project proposed herein will build directly upon our work in the P20 grant and will set the stage for the planned R01 RCT, which would be directly responsive to NCI PAR 12-275. The ultimate aim is to inform best practices in survivorship planning in community and academic cancer centers, serving diverse, including underserved minority populations, with sufficient power to detect differences between treatment groups.

OUTLINE: Patients and their caregivers participate in an upfront survivorship care planning session.

Patients and their caregivers meet with the Survivorship Nurse Practitioner (NP) at the VICC or the Nurse Navigator (NN) at MMC during an initial survivorship care planning session (30 minutes total) to identify resources that may be needed during and following therapy. The patient and their caregiver then meet together with the NP or NN (60 minutes total) to discuss the planned therapy, the expected course of recovery and recommendations for follow-up, and are provided with a preliminary survivorship care plan (SCP). Caregivers also receive the National Cancer Institute publication, "When Someone You Love is Being Treated for Cancer". Patients and their caregivers proceed with therapy. At the end of therapy, patients and their caregivers schedule a one-hour visit with the NP or NN for a booster survivorship care planning session (SCPS). At this booster session, they will review the questionnaires and receive an individualized final SCPS and the "REACH for Survivorship" handbook.

After completion of treatment for cancer, patients and their caregivers complete follow up assessments at the end of treatment and again two months after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed adult cancer patients from VICC and MMC
* Caregiver of enrolled newly diagnosed adult cancer patients from VICC and MMC
* No prior history of malignancy other than non-melanoma skin cancer
* Planned treatment for stages I - III cancer
* Treatment expected to be completed within 12 months
* English speaking

Exclusion Criteria:

* Prior history of malignancy other than non-melanoma skin cancer
* Patients treated with surgery alone will not be included
* Patients whose treatment is expected to last more than 12 months
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2015-05; Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Patient and caregiver engagement, measured by the PHQ, IES-R, Distress Thermometer, & Effective Consumer Scale-17 & Psychosocial well-being, measured by the Patient Health Questionnaire (PHQ), Impact of Event Scale-Revised (IES-R), & Distress Thermometer | Up to 2 months following the end of therapy
  Will be compared between participants (patients and caregivers) and between those treated at VICC and MMC. Will use continuous scores on the depression, anxiety, and somatic symptom scales for the primary analyses; supplemental analyses will examine the percentage of patients above and below the recommended clinical cut-offs on these scales before and after the interventions. Will develop a regression model with the treatment group as the primary variable of interest.

SECONDARY OUTCOMES:
Adherence to National Comprehensive Cancer Network (NCCN) guidelines, as measured by chart review (patients only) | Up to 2 months following the end of therapy
  Will develop a regression model with the treatment group as the primary variable of interest.
Referral to subspecialists | Up to 2 months following the end of therapy
  Will develop a regression model with the treatment group as the primary variable of interest.
Resource utilization, as measured by the Effectiveness in Obtaining Resources Scale and the Cancer Resource Survey | Up to 2 months following the end of therapy
  Will develop a regression model with the treatment group as the primary variable of interest.
Usefulness of navigation, as measured by the Usefulness of Navigator instrument | Up to 2 months following the end of therapy
  Will develop a regression model with the treatment group as the primary variable of interest.

OTHER OUTCOMES:
Completion rates | Up to 2 months following the end of therapy
  Will be descriptive. Will develop a regression model with the treatment group as the primary variable of interest. Will conduct univariable tests of significance using chi-squared tests.
Participation rates | Up to 2 months following the end of therapy
  Will be descriptive. Will develop a regression model with the treatment group as the primary variable of interest. Will conduct univariable tests of significance using chi-squared tests.
Process assessment, as measured by process evaluation questionnaire | Up to 2 months following the end of therapy
  Will be descriptive. Will develop a regression model with the treatment group as the primary variable of interest. Will conduct univariable tests of significance using chi-squared tests.

CONTACTS AND LOCATIONS:
Overall Officials: Debra Friedman, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (2):
- United States (2):
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/